CLINICAL TRIAL: NCT05476510
Title: Comparison of the Efficacy of US-guided M-Tapa Block vs OSTAP for Postoperative Analgesia in Patients After Laparoscopic Inguinal Hernia Repair Surgery
Brief Title: M-Tapa vs OSTAP for Laparoscopic Inguinal Hernia Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 29
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Inguinal Hernia
Keywords: Laparoscopic inguinal hernia repair; Postoperative pain management; Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block; Oblique Subcostal Transversus Abdominis Plane Block
MeSH Terms: conditions — Hernia, Inguinal; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for laparoscopic inguinal hernia repair surgery will be included in the study. Patients will be randomly divided into two groups (Group M TAPA = M-TAPA group, Group OSTAP = OSTAP group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant will be blinded to the stud
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA = M-TAPA Block Group (Active Comparator): Under aseptic conditions, a high-frequency linear probe will be placed on the costochondral angle in the sagittal plane. Then the probe will be slightly angled deeply to visualize the lower view of the perichondrium. We will perform M-TAPA with total of 60 ml (30 ml for each side) of %0,25 bupivacaine.
  Interventions: Drug: Postoperative management
- Group OSTAP = OSTAP Block Group (Active Comparator): In the supine position, the transducer is placed in the subcostal region in an oblique plane, and a 15-20 cm needle is first inserted between the rectus abdominis and the transversus abdominis muscle and advanced towards the iliac crest in the interfascial plane. The block location will be confirmed with 5 ml of saline. After the block location is confirmed, a total of 30 ml + 30 ml of 0.25% bupivacaine (total of 60 ml for both sides) will be injected bilaterally.
  Interventions: Drug: Postoperative management

INTERVENTIONS:
Drug: Postoperative management — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. 100 mg tramadol will be performed for rescue analgesia.

SUMMARY:
Inguinal hernia repair is the most common of abdominal surgical procedures and is usually performed laparoscopically. Many factors play a role in the pain that develops after surgery and is generally considered to be visceral pain. Phrenic nerve irritation due to CO2 insufflation into the peritoneal cavity, abdominal distention, tissue trauma, sociocultural status, and individual factors are the factors that play a role in the occurrence of this pain.

Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block performed with ultrasound (US) is a new block that provides effective analgesia in the anterior and lateral thoracoabdominal areas, where local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and abdominal lateral wall and may be an opioid-sparing strategy with satisfactory quality recovery in patients undergoing laparoscopic surgery.

Oblique Subcostal Transversus Abdominis Plane Block (OSTAP) is one of the body blocks used especially for postoperative analgesia. OSTAP, defined by Hebbard in 2010, is a subcostal version of the Transversus abdominis plane block (TAP block), based on the injection of local anesthetic from the lower edge of the costal margin, obliquely between the obliquus externus and Transversus abdominis muscles.

This study aimed to compare the efficacy of US-guided M-TAPA block and OSTAP block for postoperative analgesia management after laparoscopic inguinal hernia repair surgery. Our primary aim is to compare postoperative pain scores (0. hour NRS), and our secondary aim is to evaluate the use of rescue analgesics (opioids), side effects associated with opioid use (allergic reaction, nausea, vomiting), and patient satisfaction (Likert scale).

DETAILED DESCRIPTION:
Inguinal hernia repair is the most common of abdominal surgical procedures and is usually performed laparoscopically. Many factors play a role in the pain that develops after surgery and is generally considered to be visceral pain. Phrenic nerve irritation due to CO2 insufflation into the peritoneal cavity, abdominal distention, tissue trauma, sociocultural status, and individual factors are the factors that play a role in the occurrence of this pain.

Postoperative pain is acute pain accompanied by an inflammatory process due to surgical trauma and gradually decreases with tissue healing. Postoperative pain is a serious problem that reduces patient comfort and delays the patient's return to work after surgery. Successful postoperative analgesia occurs in the patient due to pain; It is a known fact that it prevents many of the effects such as being unable to breathe easily and delayed mobilization.

Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block performed with ultrasound (US) is a new block that provides effective analgesia in the anterior and lateral thoracoabdominal areas, where local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral wall and may be an opioid-sparing strategy that provides a satisfactory quality improvement in patients undergoing laparoscopic surgery. M-TAPA block provides analgesia in the abdominal region at the T5-T11 level. Sonoanatomy is easy to visualize and the spread of local anesthetic can be easily seen under US guidance. With the cephalocaudal spread of the local anesthetic solution, analgesia occurs in several dermatomes. In the literature, there are studies investigating the effectiveness of M-TAPA block for postoperative pain management in bariatric surgery.

Oblique Subcostal Transversus Abdominis Plane Block (OSTAP) is one of the body blocks used especially for postoperative analgesia. OSTAP, which Hebbard defined in 2010, is a subcostal version of the Transversus abdominis plane block (TAP block) and is based on the injection of local anesthetic from the lower edge of the costal margin, obliquely between the obliquus externus and Transversus abdominis muscles. OSTAP; Although it is frequently used in laparoscopic abdominal surgery, it is a very difficult block to implement. There are studies reporting that it provides successful analgesia after various abdominal surgeries.

This study aimed to compare the efficacy of US-guided M-TAPA block and OSTAP block for postoperative analgesia management after laparoscopic inguinal hernia repair surgery. Our primary aim is to compare postoperative pain scores (0. hour NRS), and our secondary aim is to evaluate the use of rescue analgesics (opioids), the side effects associated with opioid use (allergic reaction, nausea, vomiting), and patient satisfaction (Likert scale).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic inguinal hernia repair surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* anticoagulant treatment
* local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores (Numerical Ratin Scala; 0=no pain, 10=the worst pain felt) | Postoperative 24 hours period
  NRS at postoperative 0th hour

SECONDARY OUTCOMES:
The use of rescue analgesia | Postoperative 24 hours period
  Tramodol using
Patient satisfaction scale (seven item likert scale; extremely dissatisfied, mostly dissatisfied, somewhat dissatisfied, neutral, somewhat satisfied, mostly satisfied, extremely satisfied) | Postoperative 24 hours period
  This scoring system includes evaluating the satisfaction level of patient

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940
- [Background] Aikawa K, Tanaka N, Morimoto Y. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides a sufficient postoperative analgesia for laparoscopic sleeve gastrectomy. J Clin Anesth. 2020 Feb;59:44-45. doi: 10.1016/j.jclinane.2019.06.020. Epub 2019 Jun 15. No abstract available. PMID 31212124
- [Background] Ciftci B, Alici HA, Ansen G, Sakul BU, Tulgar S. Cadaveric investigation of the spread of the thoracoabdominal nerve block using the perichondral and modified perichondral approaches. Korean J Anesthesiol. 2022 Aug;75(4):357-359. doi: 10.4097/kja.22137. Epub 2022 Apr 26. No abstract available. PMID 35468713